CLINICAL TRIAL: NCT03678454
Title: Prospective Registry of Iclusig® (Ponatinib) Used in Clinical Practice for the Treatment of Patients With Chronic Myeloid Leukemia or Ph+ Acute Lymphoblastic Leukemia in Belgium
Brief Title: Iclusig® (Ponatinib) in Clinical Practice for the Treatment of Chronic Myeloid Leukemia or Ph+ Acute Lymphoblastic Leukemia in Belgium
Status: Completed | Type: Observational
Sponsor: Incyte Biosciences Benelux (Industry)
Responsible Party: Sponsor
Organization: Incyte Corporation (Industry)
Other Study IDs: Incyte-30006
Record Dates: First submitted 2018-09-18; First posted 2018-09-19 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Chronic Myeloid Leukemia; CML; Philadelphia Chromosome-positive Acute Lymphoblastic Leukemia; Ph+ ALL
Keywords: Chronic myeloid leukemia; Philadelphia chromosome positive acute lymphoblastic leukemia; Iclusig®; ponatinib
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective registry is initiated to follow up on the use of Iclusig® in patients with CML or Ph+ ALL in routine practice in Belgium.

ELIGIBILITY:
Inclusion Criteria:

* Patient with confirmed diagnosis of:

  * CML (chronic, accelerated or blast phase) who is resistant or intolerant to dasatinib or nilotinib; and for whom subsequent treatment with imatinib is not clinically appropriate; or who has the T315I mutation.
  * Ph+ ALL who is resistant or intolerant to dasatinib and for whom subsequent treatment with imatinib is not clinically appropriate, or who has the T315I mutation.
* Patients on treatment with Iclusig® or prescribed for treatment with Iclusig® during the registry (treatment decisions should be taken outside the registry).
* Written informed consent obtained from the patient, if still alive (NPP participants that were still on Iclusig® treatment on 01 March 2016, but who died before the start of this registry will be included without informed consent provided that a waiver is granted by the ethics committee for inclusion of these patients).

Exclusion Criteria:

• Concurrently participating in a clinical study, at any time during the registry period, in which the patient is exposed to Iclusig® or to another investigational product/ vaccine (pharmaceutical product/ device).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population will include adult patients with CML or Ph+ ALL for whom the decision to initiate treatment with Iclusig® as per the indication in the product label has been made before entering in the registry. Approximately 25 haematology practices will be selected for participation in this registry.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-02-03 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Prescribed dose of Iclusig® in routine practice in Belgium | Up to 3 years
  Prescribed dose of Iclusig® in milligrams.

SECONDARY OUTCOMES:
Overall clinical benefit rate of Iclusig® based on response criteria for CML or Ph+ ALL in Belgium | Up to 3 years
  Includes treatment effectiveness, complete hematologic response, cytogenetic response, major molecular response.
Estimate of additional health care utilization cost | Up to 3 years
  Costs associated with the treatment of Iclusig®-related adverse events reported during the registry.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Beck, PhD, Study Director — Incyte Biosciences Benelux
Locations (19):
- Belgium (19):
  - ZNA Stuyvenberg, Antwerp
  - UZ Antwerpen, Antwerp
  - AZ Klina, Brasschaat
  - AZ St-Jan Brugge, Bruges
  - Institut Jules Bordet, Brussels
  - CHU Brugmann, Brussels
  - Hopital Erasme, Brussels
  - UZ Brussel, Brussels
  - Clinique universitaires Saint-Luc, Brussels
  - Ziekenhuis Oost Limburg (ZOL), Ghent
  - Hopital Jolimont, Haine-Saint-Paul
  - Jessa Ziekenhuis, Hasselt
  - AZ Groeninge, Kortrijk
  - UZ Leuven, Leuven
  - CHU Sart Tilman Liège, Liège
  - CHU Charleroi Vésale, Montigny-le-Tilleul
  - AZ Turnhout St-Elisabeth, Turnhout
  - CHR La Tourelle, Verviers
  - CHU/UCL Namur Mont-Godinne, Yvoir

REFERENCES:
- [Derived] Devos T, Deeren D, Theunissen K, Selleslag D, Bailly B, Havelange V, Lewalle P, Meers S, Benghiat FS, Gadisseur A, Granacher N, Vanstraelen G, Vellemans H, Becker A, Janssen M, Vrelust I, Lejeune M, Van de Velde A, Triffet A, Beck M, Sebti H, Mazure D. Real-world outcomes in patients with Philadelphia chromosome-positive acute lymphoblastic leukemia or chronic myeloid leukemia treated with ponatinib - final 6-year results from a Belgian registry. Hematology. 2025 Dec;30(1):2534196. doi: 10.1080/16078454.2025.2534196. Epub 2025 Aug 14. PMID 40811042